CLINICAL TRIAL: NCT04517682
Title: SARS -CoV-2 Detection in Saliva Samples: A Test Validation Protocol
Brief Title: COVID-19 and SARS-CoV-2 Detection in Saliva
Status: Completed | Type: Observational
Sponsor: Ambry Genetics (Industry)
Collaborators: The Saratoga Hospital (Unknown); St. Joseph Hospital of Orange (Other); Crozer-Keystone Health System (Other)
Responsible Party: Sponsor
Other Study IDs: COV_20_001
Record Dates: First submitted 2020-05-19; First posted 2020-08-18 (Actual); Last update posted 2022-03-07 (Actual); Status verified 2022-03

CONDITIONS: RNA Virus Infections
Keywords: Detection
MeSH Terms: conditions — RNA Virus Infections | interventions — COVID-19 Nucleic Acid Testing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — De-identified samples may be retained for 90 days.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Positive for SARS-CoV-2: Individuals who are symptomatic for COVID 19 disease, at high risk of infection or part of a screening program will provide samples for analysis which may reveal a positive result.
  Interventions: Diagnostic Test: RT-PCR
- Negative for SARS-CoV-2: Individuals who are symptomatic for COVID 19 disease, at high risk of infection or part of a screening program will provide samples for analysis which may reveal a negative result.
  Interventions: Diagnostic Test: RT-PCR

INTERVENTIONS:
Diagnostic Test: RT-PCR — The RT-PCR assay will be performed on paired nasopharyngeal and saliva samples

SUMMARY:
This study aims to validate the use of human saliva as a substrate for an assay to detect SARS-CoV-2 and define accuracy, analytical sensitivity and specificity of the TaqPath RT-PCR test.

DETAILED DESCRIPTION:
Investigators will carry out validation of a laboratory assay to detect SARS-CoV-2 nucleic acids in human saliva samples. Data for the validation will include the test results from standard nasopharyngeal (NP) swabs (controls) AND matched saliva samples (experimental group) of individuals who are either known to be infected or at high risk of being infected. Investigators hypothesize that the performance of an assay designed specifically for saliva will not perform differently, as defined by a predetermined margin, from the standard assay performed on NP and other respiratory samples

ELIGIBILITY:
Inclusion Criteria:

* Reads and understands English or Spanish
* Willing and able to provide consent
* Diagnosed with COVID-19 or at high risk of disease based on objective criteria

Exclusion Criteria:

* Unwilling or unable to provide consent.
* Pregnant female

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The population will be comprised of individuals age 18 years or older who are willing and able to provide verbal consent to provide a saliva sample AND a NP swab. The number of participants required is estimated to be 300 individuals whose infection status is unknown or 50 infection positive individuals and 50 infection negative individuals. The population will generally be symptomatic for, or at high risk of COVID-19 disease by criteria set forth in local testing sites. In addition, investigators will collect paired NP swabs and saliva from an equivalent size cohort of individuals known or suspected to NOT be infected with SARS-CoV-2.
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2020-05-21 (Actual); Primary Completion 2021-03-16 (Actual); Study Completion 2021-08-05 (Actual)

PRIMARY OUTCOMES:
Detection of COVID-19 SARs-CoV-2 in saliva samples versus nasopharyngeal samples | up to 7 days
  TaqPath RT-PCR assay performed on saliva compared to TaqPath RT-PCR performed on nasopharyngeal samples for assay accuracy, concordance, reproducibility/precision, analytical sensitivity and analytical specificity.

OTHER OUTCOMES:
Reason for testing | Baseline
  Participants may be recruited from individuals presenting for various indications for testing including; followup testing after previous positive result, at risk healthcare worker, exposure to known positive or symptomatic, public facing worker or workplace hazards, employee based screening.
Current symptom status | Baseline
  Participant is symptomatic or asymptomatic
Current symptoms | Baseline
  Participant reports one or more of the following symptoms at baseline. Cough, Shortness of breath or difficulty breathing, fever, chills, muscle pain, sore throat, new loss of taste or smell, any nausea, vomiting or diarrhea.
Prior symptoms | Baseline
  Participant reports one or more of the following symptoms at baseline. Cough, Shortness of breath or difficulty breathing, fever, chills, muscle pain, sore throat, new loss of taste or smell, any nausea, vomiting or diarrhea.
Date of first symptom or number of days since first symptom. | Baseline
  Participant reports date of first symptom or number of days since first symptom.
Previous test for COVID-19 and date of test. | Baseline
  Participant reported result (positive, negative, inconclusive) of previous test for COVID-19 and date of test .

CONTACTS AND LOCATIONS:
Overall Officials: Brigette Tippin Davis, PhD, Principal Investigator — Ambry Genetics
Locations (1):
- Ambry Genetics, Aliso Viejo, California, United States

IPD SHARING:
Plan to Share IPD: No